CLINICAL TRIAL: NCT00089726
Title: A Phase II Randomized Study of GM-CSF Gene-Modified Autologous Tumor Vaccine (CG8123) With and Without Low-Dose Cyclophosphamide in Advanced Stage Non-Small Cell Lung Cancer
Brief Title: A Cancer Vaccine (CG8123) Given With and Without Cyclophosphamide for Advanced Stage Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0031
Record Dates: First submitted 2004-08-11; First posted 2004-08-12 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Lung Cancer; Carcinoma, Non-Small-Cell Lung
Keywords: cancer vaccine; NSCLC; immunotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide

INTERVENTIONS:
Biological: CG8123
Drug: Cyclophosphamide

SUMMARY:
The main purpose of this research study is to determine if a vaccine made from a patient's lung cancer tumor cells will be effective in making the cancer shrink or disappear. The vaccine will be given by itself to some patients, while other patients will get the vaccine with cyclophosphamide (a type of chemotherapy). Studies in animals and other cancer vaccine trials suggest that cyclophosphamide may make tumor vaccines more potent. This study will try to determine if vaccine given with or without this chemotherapy is effective in destroying lung cancer cells. Additionally, the study will collect information on vaccine safety, both with and without chemotherapy, and whether the vaccine improves lung cancer-related symptoms (e.g., shortness of breath).

Tumors from surgical resection will be processed and made into a vaccine. Prior to treatment, patients will be randomized equally to one of two treatment groups, Cohort A and Cohort B. Patients in Cohort A will be treated with CG8123 vaccine only and patients in Cohort B will be treated with CG8123 vaccine plus a single dose of cyclophosphamide administered one day prior to the first, third, and fifth vaccine treatments. Patients will receive intradermal (beneath the skin) vaccine injections every two weeks for up to eight weeks, for a total of up to five vaccine treatments. The duration of this study, including active follow up, is approximately two years. After this, patients will be followed-up yearly for a total of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Suspicious diagnosis of or histologically- confirmed stage IIIB or IV non small-cell lung cancer
* Accessible and adequate tumor source for vaccine production.
* Tumor source for vaccine production must be accessible by a minor surgical procedure performed under local or regional anesthesia (e.g. lymph node or soft tissue mass or malignant pleural effusion)
* Measurable disease to evaluate following tumor procurement
* Limited metastatic tumor burden
* Life expectancy at least 4 months
* ECOG Performance Status 0 - 1

Exclusion Criteria:

* Active and/or untreated brain metastases
* Active or impending spinal cord compression
* Active auto-immune disease or treatment with immunosuppressants
* Decompensated congestive heart failure or recent significant cardiac event
* Coexisting malignancies
* Significant or uncontrolled medical problems or laboratory abnormalities that might increase the risk of surgical complications or vaccine treatment
* Previous treatment with gene therapy (including any adenoviral-based therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-03; Study Completion 2006-01 (Actual)

REFERENCES:
- See also: Related Info — http://www.cellgenesys.com